CLINICAL TRIAL: NCT06616961
Title: Efficacy and Safety of Semaglutide in Weight Reduction in Overweight or Obese Bangladeshi Adults With or Without Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of Semaglutide for Weight Loss in Overweight or Obese Adults in Bangladesh With or Without Type 2 Diabetes Mellitus
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Popular Medical College Hospital (Other)
Collaborators: Pi Research and Development Center, Bangladesh (Unknown); Incepta Pharmaceuticals Ltd (Industry)
Responsible Party: Principal Investigator, Prof. Dr Quazi Tarikul Islam, Professor, Department of Medicine, Popular Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: No.BSMMU/2024/7591
Record Dates: First submitted 2024-09-21; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Obesity; Type 2 Diabetes Mellitus (T2DM)
Keywords: Semaglutide; Obesity; Overweight; Type 2 Diabetes Mellitus (T2DM); Weight Loss; Efficacy; Safety; Bangladesh
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Overweight; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Semaglutide (Experimental): This study features a single treatment arm where participants receive semaglutide (Fitaro) for weight management. Administered subcutaneously once weekly, the treatment begins at 0.25 mg and escalates to a maximum of 2.4 mg over 16 weeks based on individual response and tolerance. Participants include overweight or obese adults aged 18 and older, with or without Type 2 Diabetes Mellitus (T2DM). The primary focus is to assess the efficacy and safety of semaglutide in achieving significant weight loss, while also evaluating its impact on metabolic parameters like body mass index (BMI), waist circumference, blood glucose levels, and overall quality of life. Alongside medication, participants will receive lifestyle counseling to encourage dietary adjustments and increased physical activity. Regular follow-up assessments will be conducted to monitor weight loss progress, metabolic health, and any treatment-related adverse events throughout the study duration.
  Interventions: Drug: Semaglutide Pen

INTERVENTIONS:
Drug: Semaglutide Pen — In this study, the intervention involves administering semaglutide (Fitaro) to participants for weight management. The treatment protocol includes the following steps:
  Initial Dose: Participants will start with a subcutaneous injection of semaglutide at a dose of 0.25 mg once weekly for the first four weeks to allow for tolerance and adjustment.
  Dose Escalation: After the initial period, the dose will be increased at four-week intervals as follows:
  Week 5: Increase to 0.5 mg Week 9: Increase to 1 mg Week 13: Increase to 1.7 mg Week 17: Increase to a maximum dose of 2.4 mg, if necessary, based on individual weight loss response and tolerability.
  Other Names: Semaglutide Pen without ADA

SUMMARY:
The goal of this clinical trial is to learn if semaglutide can help with weight loss in overweight or obese adults in Bangladesh. The study will also look at how safe semaglutide is for these participants. The main questions to answers are given below:

Does semaglutide help participants lose weight after 26 weeks? What changes occur in health measures like blood sugar and quality of life for those taking semaglutide?

Participants will:

Receive a weekly injection of semaglutide (2.4 mg) for 26 weeks. Follow a plan that includes lifestyle changes, such as diet and physical activity.

Have their body weight, waist size, and blood sugar levels measured regularly. This study aims to provide important information on how well semaglutide works for weight loss in Bangladeshi adults, helping to find effective treatments for obesity in this population.

DETAILED DESCRIPTION:
Background and Rationale Obesity has emerged as a significant global health challenge, with its prevalence increasing rapidly across various demographics. Estimates suggest that nearly half of the world's population could be classified as overweight by the year 2030. The ramifications of this trend are profound, leading to increased risk for a variety of chronic diseases, including type 2 diabetes mellitus (T2DM), hypertension, dyslipidemia, and several cardiovascular diseases. In fact, obesity is estimated to be responsible for approximately five million deaths globally each year, with a notable mortality rate of 62.6 deaths per 100,000 individuals suffering from obesity. Although the mortality rates in low- and middle-income countries are lower than in developed regions, trends indicate a concerning increase in obesity-related mortality in these areas.

Even modest weight loss (5-10% of body weight) can lead to significant health benefits, such as slowing the progression of T2DM and reducing cardiovascular risks. Moreover, evidence indicates that weight reduction can correlate with an 18% reduction in premature mortality. Traditional weight management strategies primarily involve lifestyle modifications such as dietary changes and increased physical activity; however, many individuals find it difficult to achieve and sustain these changes.

While surgical options are available for severe cases of obesity, they come with inherent risks and complications that necessitate ongoing follow-up care. In this context, pharmacotherapy offers a valuable adjunct to lifestyle interventions, helping individuals achieve and maintain clinically relevant weight loss while potentially improving coexisting health conditions.

Currently, there are limited anti-obesity medications available; thus, there is a pressing need for more effective therapeutic options that can aid in weight maintenance and comorbidity prevention. Among the medications approved for long-term use is semaglutide, a glucagon-like peptide-1 receptor agonist initially developed for the treatment of T2DM. Recent studies have demonstrated its effectiveness in promoting weight loss, particularly in Caucasian populations.

However, existing trials primarily include participants from Europe and North America. This raises questions about the applicability of these findings in Asian populations, such as those in Bangladesh, where genetic and environmental factors can influence obesity outcomes significantly. Morphological differences exist between populations; for instance, central obesity is more prevalent among Caucasians, while subcutaneous fat accumulation is common in Asians.

In Bangladesh, semaglutide (Fitaro) is available for weight management at various doses (0.25 mg to 2.4 mg), but there is a lack of specific evidence regarding its efficacy and safety in this demographic. This study aims to fill that gap by investigating the effectiveness of semaglutide in overweight or obese individuals with or without T2DM within the Bangladeshi population.

Study Objectives and Hypothesis Research Question

* What is the role of semaglutide in managing obesity and overweight among the Bangladeshi population? Hypotheses
* Null Hypothesis: Semaglutide is not effective in managing obesity and overweight among the Bangladeshi population.
* Alternative Hypothesis: Semaglutide is effective in managing obesity and overweight among the Bangladeshi population.

Objectives

Primary Objective:

• To assess the efficacy and safety of semaglutide administered once weekly for weight loss in overweight or obese patients with or without T2DM.

Secondary Objectives:

* To evaluate the efficacy and safety of semaglutide for weight reduction in overweight or obese individuals without T2DM.
* To investigate the efficacy and safety of semaglutide for weight reduction in overweight or obese individuals with T2DM.
* To compare the efficacy and safety profiles of semaglutide between diabetic and non-diabetic obese patients.
* To examine the effects of semaglutide on metabolic conditions associated with T2DM, hypertension, dyslipidemia, and hyperuricemia.
* To assess the impact of semaglutide on quality of life in overweight or obese patients.

Methodology Study Design This study will be a single-arm experimental trial conducted in real-world settings across multiple hospitals in Bangladesh including Popular Medical College Hospital, Dhaka Medical College Hospital, Bangabandhu Sheikh Mujib Medical University, and others.

Study Population Participants will be grouped into two categories Group A: Overweight or obese patients without T2DM. Group B: Overweight or obese patients with T2DM. Sample Size Using OpenEpi software with a significance level set at 95% and a power of 90%, we estimate needing a total sample size of approximately 480 participants (240 per group) to account for a potential dropout rate of 20%.

Inclusion Criteria Both diabetic and non-diabetic participants -

* Must provide informed consent.
* Age ≥18 years.
* BMI ≥30 kg/m² or ≥25 kg/m² with related health conditions.

For those with T2DM:

* Diagnosed for at least six months prior to screening.
* HbA1c level ≤12%. Exclusion Criteria Exclusion criteria include
* Recent significant weight loss (≥5 kg) within the last month.
* Use of any anti-obesity medications within the past three months.
* Previous surgical interventions for obesity.
* Certain medical histories including pancreatitis, major depressive disorder, and uncontrolled thyroid diseases.

Intervention Treatment Allocation All participants will receive semaglutide (Fitaro) administered subcutaneously once weekly at escalating doses starting from 0.25 mg up to a maximum of 2.4 mg, based on tolerance and response.

Dose Escalation Schedule

* Weeks 0-4: Start at 0.25 mg
* Weeks 5-8: Increase to 0.5 mg
* Weeks 9-12: Increase to 1 mg
* Weeks 13-16: Increase to 1.7 mg
* Weeks 17+: Increase to maximum dose of 2.4 mg if target weight loss is not achieved.

Lifestyle Modifications Participants will receive counseling regarding dietary changes and physical activity tailored to their needs. A balanced diet focusing on whole foods, portion control, and regular exercise will be emphasized.

Outcome Measures Primary Endpoint

* Change in body weight from baseline at week 26. Secondary Endpoints
* Change in BMI
* Waist circumference
* HbA1c levels
* Fasting blood glucose levels
* Blood pressure readings
* Lipid profiles
* Serum uric acid levels
* Overall quality of life assessed through the Obesity-Specific Quality of Life instrument (OSQOL).

Data Collection and Monitoring Data will be collected using semi-structured questionnaires administered at baseline and during follow-up visits at weeks 4, 8, 12, 16, and finally at week 26.

A Data and Safety Monitoring Board (DSMB) will oversee the study integrity by reviewing safety data at regular intervals.

Statistical Analysis Plan Data will be analyzed using SPSS software applying mixed effects linear regression models for primary outcomes and appropriate statistical tests for secondary outcomes.

Ethical Considerations The study will adhere to ethical standards set forth by Bangabandhu Sheikh Mujib Medical University's Institutional Review Board. Informed consent will be obtained from all participants prior to enrollment.

Conclusion This study aims to provide critical insights into the efficacy and safety of semaglutide for weight management among Bangladeshi adults struggling with obesity or overweight issues, presenting an opportunity to enhance treatment strategies tailored to local populations.

ELIGIBILITY:
Inclusion Criteria:

-Common inclusion criteria for both diabetic and non-diabetic individuals

* Informed consent will be obtained before any trial-related activities
* Male or female, aged ≥ 18 years at the time of signing the informed consent form
* Body mass index (BMI) ≥30 kg/m2 with or without any weight-related comorbidities or ≥25-29.9 kg/m2 with the presence of at least one of the following weight-related comorbidities (treated or untreated): hypertension, dyslipidemia, obstructive sleep apnea or cardiovascular disease (more than three months) For subjects with T2DM
* Patients diagnosed with T2DM more than or equal to 180 days prior to the day of screening.
* HbA1c up to 12.0%

Exclusion Criteria:

* Common exclusion criteria for both diabetic and non-diabetic individuals Medical criteria

  * A self-reported reduction in body weight of more than 5 kg within 30 days before screening, irrespective of medical records
  * Treatment with any medication for the indication of obesity within the past 90 days before screening (eg. Orlistat, liraglutide, naltrexone/bupropion, diethylpropion, phendimetrazine, and Setmelanotide etc.)
  * Any previous obesity treatment with surgery or a weight loss device during lifetime
  * Continued treatment with other GLP-1 agonists, SGLT-2 inhibitor and/or metformin. However, if these drugs can be stopped based on the best clinical judgement of the investigator, the patient can be recruited after stopping the drug and a washout period of two weeks. In case of semaglutide (ORSEMA) the wash out period will be 10 weeks.
  * Patient taking oral or injectable steroid for other indications
  * Past history of pancreatitis
  * Diagnosed case of eating disorders eg. Bulimia nervosa
  * Patients with a previous history of suicide attempts and major depressive disorder (MDD) according to the DSM-V criteria, schizophrenia or anti-psychotic drug induced obesity
  * Patients with a personal or family history of medullary thyroid carcinoma (MTC) and/or multiple endocrine neoplasia syndrome type 2 (MEN 2)
  * Known hypersensitivity to Semaglutide or any of the product components.
  * History of recent MI (within past three months)
  * Pregnancy and lactation Laboratory criteria
  * Incidental diagnosis or Uncontrolled thyroid disease, defined as a thyroid stimulating hormone (TSH) level > 6.0 mIU/L or <0.4 mIU/L as measured by the central laboratory at screening. However, well-controlled thyroid disorder can be included if TSH<6.0 or >0.4 mIU/L.
  * Renal impairment, measured as the estimated glomerular filtration rate (eGFR) <15 ml/min/1.73 m2 For subjects without T2DM
  * HbA1c more than or equal to 48 mmol/mol (6.5%) For subjects with T2DM
  * Renal impairment, defined as an estimated glomerular filtration rate (eGFR) less than 30 mL/min/1.73 m2 (less than 60 mL/min/1.73 m2 in subjects treated with a sodium-glucose cotransporter 2 inhibitor (SGLT2i)).
  * Uncontrolled T2DM (HbA1c >12.0%) as these patients may require insulin or other anti-diabetic drug which might potentially interfere the efficacy of semaglutide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Body Weight (kg) | 26 weeks
  Measured at baseline (week 0) and at week 26, with specific targets for weight loss of 5%, 10%, 15%, and 20%.

SECONDARY OUTCOMES:
BMI (kg/m²) | 26 weeks
  Body Mass Index (BMI) is calculated using the formula: BMI=weight (kg)/height (m)2
Waist circumference (cm) | 26 weeks
  Waist circumference measures the size of a person's waist and indicates body fat distribution. To measure, find the natural waistline above the belly button, wrap a flexible measuring tape around it, and record the measurement.
HbA1C (%) | 26 weeks
  HbA1c, or glycated hemoglobin, measures average blood sugar levels over the past 3 months.
FPG (mmol/l) | 26 weeks
  Fasting blood glucose
Systolic blood pressure (mmHg) | 26 weeks
  Systolic Blood Pressure (SBP) is the pressure in your arteries when your heart beats, representing the maximum pressure during heart contraction. It is the higher number in a blood pressure reading, such as 120 in 120/80 mmHg
Diastolic blood pressure (mmHg) | 26 weeks
  Diastolic pressure is the lower number in a blood pressure reading, indicating the pressure in the arteries when the heart is at rest between beats. It reflects the minimum pressure in the arteries and is important for assessing cardiovascular health.
Total cholesterol (mg/dl) | 26 weeks
  Total cholesterol is a measure of the combined levels of cholesterol in your blood, including low-density lipoprotein (LDL), high-density lipoprotein (HDL), and very low-density lipoprotein (VLDL). It is an important indicator of heart health, as high levels can increase the risk of heart disease and stroke. Total cholesterol levels are usually measured in milligrams per deciliter (mg/dL).
Triglyceride | 26 weeks
  Triglycerides are a type of fat (lipid) found in your blood. They are used by the body for energy and are stored in fat cells. High levels of triglycerides can increase the risk of heart disease, especially when combined with low HDL (good cholesterol) or high LDL (bad cholesterol). Triglyceride levels are typically measured in milligrams per deciliter (mg/dL).
Dose alteration | 26 weeks
  Change or increment of hypoglycemic agents in patients with T2DM Reduction or increment of antihypertensive drugs in patients with hypertension
Quality of Life | 26 weeks
  The Obesity-specific Quality of Life instrument (OSQOL) evaluates four key domains: physical state, vitality, social interactions, and psychological state. This assessment is conducted over a 26-week period to gauge changes in quality of life specific to individuals with obesity. When reporting scores, it's essential to include the full scale title, along with the minimum and maximum values. For clarity, specify whether higher scores indicate a better or worse outcome, ensuring that the results provide meaningful insights into the participants' quality of life.
Safety endpoints | 26 weeks
  Adverse Events: Number of treatment-related adverse events from baseline to week 26.
  Serious Adverse Events (SAEs): Number of SAEs from baseline to week 26.

CONTACTS AND LOCATIONS:
Locations (1):
- Popular Medical College Hospital, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No